CLINICAL TRIAL: NCT03857555
Title: Causes of Peripheral Hypotonia in Children Attending Assiut University Children Hospital
Brief Title: Causes of Peripheral Hypotonia in Assiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Azza Abouzeid Zaki, principle investigator, Assiut University
Other Study IDs: COPHIAUCH
Record Dates: First submitted 2019-02-14; First posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Infant Floppy
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypotonia is a common manifestation in infants and children.It includes several clinical conditions that do not always lead to a favorable outcome .Thus, it is important to make early diagnosis to decide on the treatment and follow up of these cases. Hypotonia is a state of low muscle tone (The amount of tension or resistance to stretch on a muscle), often pointing to reduced muscle strength.

Hypotonia is not a specific medical disorder, but a potential manifestation of several diseases and disorders, that affect motor nerve control by the brain or muscle strength.

DETAILED DESCRIPTION:
Criteria of peripheral hypotonia are : absent or depressed tendon reflexes , failure of movements on postural reflexes ,fasciculation with or without muscle atrophy .A sequential scheme of localization would begin with the anterior horn cell (AHC), and progress to the peripheral nerve , neuromuscular junction (NMJ) and the muscle itself.

Electroneuromyography (ENMG) provides useful information on many neuromuscular diseases. In addition nerve conduction study is also helpful to identify the most common peripheral disorders causing hypotonia in these children.

The initial approach to hypotonia is to determine whether the problem is due to central or peripheral origin.This is of crucial importance when forming a plan for diagnostic investigations and management.

Many muscle diseases share common clinical features that may lead to laboratory diagnosis by using enzyme levels that are affected in some of these diseases(e.g creatine phosphokinase ). However the use of serum creatine phosphokinase level may not possibly differentiate between various muscle diseases . The selective involvement of certain muscles is a key to the diagnosis of muscle disease].

High resolution ultrasound allows visualization of the muscle, nerve and adjacent structures and can offer real-time information regarding neuromuscular diseases. It can be used as a helping tool to electrodiagnosis with estimation of the serum creatine phosphokinase levels of these cases.

The aim of this work :is to give a profile of the causes of peripheral hypotonia in infant and children attending Assiut University Children Hospital during one year of the study .

Besides full clinical assessment of the cases including birth history , developmental history, age, sex, and duration of illness as well as age of onset of observed weakness will be recorded. Full neurological examination will be done in all cases .Cases will have serum creatine phosphokinase levels, electromyography and nerve conduction studies done as indicated.Cases will also have real time muscle ultrasonography done.

* Our results will be compared with the results obtained by other investigators .
* Statistical analysis : correlation studies will be done between the various methods of investigations used .Chi2 test will be used to indicate the prevalence of the various causes of hypotonia found in the study .

ELIGIBILITY:
Inclusion Criteria:

* all infant and children with peripheral hypotonia

Exclusion Criteria:

* central causes of hypotonia

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will be conducted in the neuro-pediatric clinic at Assiut University Hospital after approval from the ethical review board.Tthirty five infant and children with peripheral hypotonia will be evaluated to reach a diagnosis
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
To detect the role of combin- ing clinical and radiological assessments in the diagnosis of muscle diseases and the possibility of using muscle ultrasound as a screening tool when muscle diseases are suspected. | 30 minutes,
  Muscles ultrasounds will perform using Phillips HD15000, brand ATL,model HTI 5000,and Origin USA linear probe 5_12MHz.The probe will use in a transverse plane,perpendicular to the long axis of the muscle.The muscle will examine through its whole length dynamically inspect for any spontaneous activity at rest. The following muscles will be inspected :1.anterior thigh:rectus femoris,vastus intermedius,lateral is and medial is,sartorius, and gracilis,2.posterior thigh:adductors,biceps femoris,semitendinous, semimembranosus, (c) leg:tepialis anterior,peronii, and gastrocnemius soleus.
  We will employ a visual grading system to detect whether the muscles affected. Normal muscle appears with low echo_intensity divided by ecchogenic perimysium and connective tissue with speckled appearance in the transverse plane.The muscle will be considered abnormal if it shows increase ecchogenicity, lost its striation, or show change in muscle bulk.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Helmy H, Aboumousa A, Abdelmagied A, Alsayyad A, Nasr SA. The role of muscle ultrasound in helping the clinical diagnosis of muscle diseases. Egypt J Neurol Psychiatr Neurosurg. 2018;54(1):29. doi: 10.1186/s41983-018-0039-6. Epub 2018 Nov 1. PMID 30459502
- [Result] Cetin E, Cuisset JM, Tiffreau V, Vallee L, Hurtevent JF, Thevenon A. The value of electromyography in the aetiological diagnosis of hypotonia in infants and toddlers. Ann Phys Rehabil Med. 2009 Sep-Oct;52(7-8):546-55. doi: 10.1016/j.rehab.2009.06.004. Epub 2009 Aug 18. English, French. PMID 19713169